CLINICAL TRIAL: NCT04231422
Title: A Proof of Concept Top Evaluate a Novel Penile Lengthening Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Judson Brandeis (Industry)
Responsible Party: Sponsor-Investigator, Judson Brandeis, Principal Investigator, BrandeisMD
Organization: BrandeisMD (Industry)
Other Study IDs: BRAND-003
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Penile Elongation
Keywords: platelet-rich plasma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment Group: Monthly intracavernosal platelet-rich plasma injection + daily physical manipulation.
  Interventions: Combination Product: Platelet-rich plasma

INTERVENTIONS:
Combination Product: Platelet-rich plasma — 12mL of platelet-rich plasma injected into cavernosal bodies bilaterally

SUMMARY:
The objective of this study is to examine and quantify the efficacy and safety of a new treatment protocol using platelet-rich plasma for penile length enhancement.

ELIGIBILITY:
Inclusion Criteria:

1. Stretched penile length between 3.5 - 8.0 in
2. Age 20-55 years of age
3. Desire penile length elongation
4. Willing to complete all aspects of combined treatment plan
5. Able to measure erect penile length and mid-shaft girth at 1-month intervals
6. Judged to be in good health based on medical history, physical exam, and laboratory profile
7. Is willing and able to cooperate with the requirement of the study (e.g. completion of all planned study visits)

Exclusion Criteria:

1. No prior surgical Peyronie's disease treatment
2. No chordee with or without hypospadias
3. No infiltration by benign or malignant mass
4. No active STD
5. No infiltration by an infectious agent such as lymphogranuloma venereum
6. No uncontrolled psychiatric conditions
7. No uncontrolled neurologic conditions
8. No other uncontrolled medical conditions such as HTN or DM
9. No history of spontaneous priapism
10. Is unable to safely use the study devices as determined by the principal investigator
11. No thrombosis of the dorsal penile artery or vein
12. No known history of coagulation disorder
13. No known history of stroke, bleeding, or another significant medical conditional which the investigator deems makes the subject unsuitable for enrollment in the study
14. Testosterone level lower than 500

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study participants comprised of men with a desire for penile elongation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-05-12 (Estimated); Study Completion 2021-07-12 (Estimated)

PRIMARY OUTCOMES:
Stretched penile length | baseline to six months
  Change in length of stretched, flaccid penile length

SECONDARY OUTCOMES:
SHIM Score | baseline to six months
  Change in erectile function
BDD-YBOCS | baseline to six months
  Change in body dysmorphia scale
Safety Measurement | baseline to six months
  Incidence of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Judson Brandeis, MD, Principal Investigator — BrandeisMD
Locations (1):
- BrandeisMD, San Ramon, California, United States

IPD SHARING:
Plan to Share IPD: Undecided